CLINICAL TRIAL: NCT02497378
Title: A Phase 1b Study of JNJ-54767414 (Daratumumab) in Combination With Bortezomib and Dexamethasone (D-Vd) in Japanese Patients With Relapsed or Refractory Multiple Myeloma (MM)
Brief Title: A Study of JNJ-54767414 (Daratumumab) in Combination With Bortezomib and Dexamethasone (D-Vd) in Japanese Participants With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR107666; 54767414MMY1005 (Other: Janssen Pharmaceutical K.K.)
Record Dates: First submitted 2015-07-10; First posted 2015-07-14 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Daratumumab; JNJ-54767414; Bortezomib; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- JNJ-54767414 (Daratumumab) +Bortezomib+Dexamethasone (Experimental): Participants will be administered JNJ-54767414 (daratumumab) intravenously at a dose of 16 milligram per kilogram (mg/kg) weekly for the first 3 cycles, then on Day 1 of Cycles 4-8 (every 3 weeks), and then on Day 1 of subsequent cycles (every 4 weeks), First 8 Cycles are 21-day cycles; Cycles 9 and onwards are 28-day cycles. Bortezomib at a dose of 1.3 milligram per meter square (mg/m^2) subcutaneously (SC) on Days 1, 4, 8 and 11 of each 21-day cycle for 8 treatment cycles and Dexamethasone orally at 20 mg on Day 1, 2, 4, 5, 8, 9, 11 and 12 of the first 8 bortezomib treatment cycles.
  Interventions: Drug: JNJ-54767414 (Daratumumab); Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: JNJ-54767414 (Daratumumab) — JNJ-54767414 (Daratumumab) will be administered as an Intravenous (IV) infusion at a dose of 16 milligram per kilogram (mg/kg) weekly for the first 3 cycles, on Day 1 of Cycles 4-8 (every 3 weeks), and then on Day 1 of subsequent cycles (every 4 weeks). First 8 Cycles are 21-day cycles; Cycles 9 and onwards are 28-day cycles.
Drug: Bortezomib — Bortezomib will be administered at a dose of 1.3 mg/m^2 subcutaneously (SC) on Day 1, 4, 8 and 11 of each 21-day cycle. Eight Bortezomib treatment cycles are to be administered.
  Other Names: VELCADE
Drug: Dexamethasone — Dexamethasone will be administered orally at 20 mg on Day 1, 2, 4, 5, 8, 9, 11 and 12 of the first 8 bortezomib treatment cycles (except for Cycles 1-3). In Cycles 1-3, participants receive dexamethasone 20 mg on days 1, 2, 4, 5, 8, 9, 11, 12 and 15. During weeks when the participants receives an infusion of daratumumab, dexamethasone will be administered at a dose of 20 mg IV or orally (PO) (only if IV is not available) before the daratumumab infusion as preinfusion medication.

SUMMARY:
The purpose of this study is to evaluate the tolerability and safety of JNJ-54767414 (daratumumab) in Combination With Bortezomib and Dexamethasone (D-Vd) in Japanese participants with relapsed (the return of a medical problem) or refractory (not responding to treatment) multiple myeloma.

DETAILED DESCRIPTION:
This is an open-label (all participants and study personnel will know the identity of the study treatments) and multicenter (study conducted at multiple sites) study in Japanese participants. The study will include a Screening Phase (21 days prior to Cycle 1 Day 1); open-label treatment phase (from Cycle 1 Day 1 until study treatment discontinuation, disease progression, unacceptable toxicity, or other reasons), and a Follow-up Phase. Bortezomib and Dexamethasone will be administered along with JNJ-54767414 for first 8 treatment cycles. Follow-up Phase begins immediately following the End-of-Treatment Visit, and will continue until 8 weeks after last study treatment, death, loss to follow-up, consent withdrawal for study participation, or study end, whichever occurs first. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants proven to have symptomatic (having symptoms) multiple myeloma (MM) according the International Myeloma Working Group (IMWG) diagnostic criteria
* Participant must have documented MM as defined by following criteria: Monoclonal plasma cells in the bone marrow 10 percent (%), or presence of a biopsy-proven plasmacytoma at some point in their disease history, disease measurements: a) Serum M-protein greater than or equal to (>=) 1 gram per deciliter (g/dL) (>=10 gram per liter [g/L]) b) Serum immunoglobulin A [IgA] M-protein >= 0.5 g/dL); c) Urine M-protein >=200 milligram per 24 hour (mg/24 h); d) Serum immunoglobulin free light chain >=10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio
* Participant must have received at least 1 prior line of therapy for MM
* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Participant must have achieved a response (partial response [PR] or better based on investigator's determination of response by the IMWG criteria) to at least 1 prior regimen

Exclusion Criteria:

* Participant has received daratumumab or other anti-cluster of differentiation 38 (anti-CD38) therapies previously
* Is refractory to bortezomib or another PI, like ixazomib and carfilzomib (had progression of disease while receiving bortezomib therapy or within 60 days of ending bortezomib therapy or another PI therapy, like ixazomib and carfilzomib
* Is intolerant to bortezomib (ie, discontinued due to any adverse event while on bortezomib treatment)
* Has received anti-myeloma treatment within 2 weeks or 5 pharmacokinetic half-lives of the treatment, whichever is longer, before the date of daratumumab first administration. The only exception is emergency use of a short course of corticosteroids (equivalent of dexamethasone 40 milligram per day [mg/day] for a maximum of 4 days) before treatment. A list of anti-myeloma treatments with the corresponding pharmacokinetic half-lives is provided in the Site Investigational Product Procedures Manual (IPPM)
* Has a history of malignancy (other than multiple myeloma) within 3 years before the date of daratumumab first administration
* Has any concurrent medical condition or disease (eg, active systemic infection, pulmonary impairment) that is likely to interfere with study procedures

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Approximately 2 years
  An AE was any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

SECONDARY OUTCOMES:
Minimum Observed Serum Concentration (Cmin) of JNJ-54767414 (Daratumumab) | Approximately 2 years
  The Cmin is the maximum observed serum concentration of JNJ-54767414.
Maximum Observed Serum Concentration (Cmax) of JNJ-54767414 (Daratumumab) | Approximately 2 years
  The Cmax is the maximum observed serum concentration of JNJ-54767414.
Serum Concentration of JNJ-54767414 (Daratumumab) Antibodies | Approximately 2 years
  Serum levels of antibodies to Daratumumab for evaluation of potential immunogenicity.
Percentage of Participants With Overall Response Rate (ORR) | Approximately 2 years
  Overall response rate is defined as the percentage of participants who achieve complete response or partial response according to the International Myeloma Working Group criteria, during or after study treatment.
Percentage of Participants with Complete Response (CR) or better | Approximately 2 years
  CR is Defined as the proportion of Participants achieving CR (including sCR) according to the IMWG criteria.
Percentage of Participants with a Very Good Partial Response (VGPR) or better | Approximately 2 years
  VGPR is defined as a greater than 90% reduction in serum myeloma protein (M-protein) plus urine myeloma protein less than 100 milligram (mg) per 24 hours.
Time to Response | Approximately 2 years
  Time to response is defined as the time from the date of first dose of study treatment to the date of the first documentation of observed response (CR or PR).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (5):
- Japan (5):
  - Hiroshima
  - Hitachi
  - Nagoya
  - Shibuya City
  - Tachikawa

REFERENCES:
- [Derived] Iida S, Ichinohe T, Shinagawa A, Suzuki K, Takezako N, Aoki M. Safety and efficacy of daratumumab in combination with bortezomib and dexamethasone in Japanese patients with relapsed or refractory multiple myeloma. Int J Hematol. 2018 Apr;107(4):460-467. doi: 10.1007/s12185-017-2390-2. Epub 2017 Dec 19. PMID 29260507
- See also: A Phase 1b Study of JNJ-54767414 (Daratumumab) in Combination With Bortezomib and Dexamethasone (D-Vd) in Japanese Patients With Relapsed or Refractory Multiple Myeloma (MM) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR107666&attachmentIdentifier=4f56a255-b7e2-4ed1-b927-a68e44a5d4fd&fileName=CR107666_CSR.pdf&versionIdentifier=